CLINICAL TRIAL: NCT00983515
Title: A One-Directional, Open-label Drug Interaction Study to Investigate the Effects of Multiple-Dose Ritonavir on Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Between Colchicine and Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice president, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1013
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Colchicine; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): -baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Ritonavir (Experimental): -colchicine pharmacokinetics in presence of steady-state ritonavir
  Interventions: Drug: Ritonavir; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of colchicine 0.6 mg administered alone at 7:00 a.m. on Day 1 after an overnight fast of at least 10 hours.
  Other Names: COLCRYS™
  Arms: Colchicine alone
Drug: Ritonavir — One 100 mg ritonavir capsule administered twice daily at 7:00 a.m. and 7:00 p.m. on Days 15 to 18 without regard to meals, then along with colchicine at 7:00 a.m. on Day 19 after an overnight fast of at least 10 hours; final dose of 100 mg ritonavir administered at 7:00 p.m. on Day 19
  Other Names: Norvir® Capsules USP, 100 mg (Abbott Laboratories)
  Arms: Colchicine with Ritonavir
Drug: Colchicine — A single dose of colchicine 0.6 mg administered along with ritonavir at 7:00 a.m. on Day 19
  Arms: Colchicine with Ritonavir

SUMMARY:
Ritonavir is a potent inhibitor of CYP3A4, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of ritonavir on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Ritonavir is a potent inhibitor of CYP3A4, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of ritonavir on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period. After a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given a single oral dose of colchicine (1 x 0.6 mg tablet) on Day 1. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis on Days 2-5. After a 14 day washout period, on study Days 15-18, subjects will return to the clinic daily for non-confined dosing of ritonavir (1 x 100 mg capsule) every 12 hours. Administered ritonavir doses on these days will not necessarily be in a fasted state. On Day 15, after taking the first dose of ritonavir, subjects will remain in the clinic for observation for 1 hour post-dose administration. On day 19 after a fast of at least 10 hours, a single dose of colchicine (1 x 0.6 mg tablet) and ritonavir (1 x 100 mg capsule) will be co-administered to all study participants. Fasting will continue for 4 hours following the co-administered doses of ritonavir and colchicine. All participants will be confined to the clinic for dosing and 24-hour blood sampling at times sufficient to adequately determine the pharmacokinetics of colchicine. Blood sampling will continue on a non-confined basis on Days 20-23. The final dose of ritonavir (1 x 100 mg capsule) will be administered to subjects the evening of Day 19, in a non-fasting state. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (blood pressure and pulse) will be measured prior to dosing and at 1, 2, and 3 hours following drug administration on Days 1, 15 and 19 to coincide with peak plasma concentrations of both colchicine and ritonavir. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive.

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, hyperlipidemia, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, East Grand Forks, Minnesota, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, male and female volunteers, consisting of members from the community at large, were enrolled in the study.
Pre-assignment Details: 48 subjects were screened, 11 were screen failures, 7 had schedule conflicts, 6 were not needed
Groups:
- Colchicine Alone / With Ritonavir (at Steady-state): [All subjects received each of the study treatments.] On Day 1, each subject received one colchicine 0.6 mg tablet at 7:00 a.m. after an overnight fast of at least 10 hours, followed by a washout period of 14 days. On Days 15 to 18, each subject received one 100 mg ritonavir capsule twice daily at 7:00 a.m. and 7:00 p.m. without regards to meals. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one 100 mg ritonavir capsule at 7:00 a.m. after an overnight fast. A final dose of ritonavir was administered at 7:00 p.m. that evening.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Ritonavir (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Ritonavir (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: Ritonavir Alone
Arm/Group | Colchicine Alone / With Ritonavir (at Steady-state)
Started | 24
Completed | 18
Not Completed | 6
Not completed — liver panel out of range | 6
Period: Colchicine With Ritonavir
Arm/Group | Colchicine Alone / With Ritonavir (at Steady-state)
Started | 18
Completed | 17 (pharmacokinetic data included since parameters could be estimated for both dosing conditions)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Ritonavir (at Steady-state)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45 years old
  Participants
    <=18 years | 5
    Between 18 and 65 years | 19
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn within 1 hour prior to colchicine dosing (0 hour) on Days 1 and 19, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours after colchicine dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: On Day 1, each subject received one 0.6 mg colchicine tablet at 7:00 a.m. after an overnight fast of at least 10 hours, followed by a washout period of 14 days.
- Colchicine With Ritonavir (at Steady-state): On Days 15 to 18, each subject received one 100 mg ritonavir capsule twice daily at 7:00 a.m. and 7:00 p.m. without regards to meals. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one 100 mg ritonavir capsule at 7:00 a.m. after an overnight fast. A final dose of ritonavir was administered at 7:00 p.m. that evening.
Arm/Group | Colchicine Alone | Colchicine With Ritonavir (at Steady-state)
Number analyzed (Participants) | 18 | 18
pg/mL | 1,869.50 (526.94) | 4,993.06 (1,257.07)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Ritonavir (at Steady-state)
Number analyzed (Participants) | 18 | 18
pg-hr/mL | 8,412.04 (3,992.34) | 29,048.45 (8,935.10)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Ritonavir (at Steady-state)
Number analyzed (Participants) | 18 | 18
pg-hr/mL | 10,410.73 (4,734.38) | 35,276.22 (10,508.55)

ADVERSE EVENTS:
Groups:
- Ritonavir Alone: On Days 15 to 18, each subject received one 100 mg ritonavir capsule twice daily at 7:00 a.m. and 7:00 p.m. without regards to meals.
- Colchicine With Steady-state Ritonavir: On Day 19, each subject received both one 0.6 mg colchicine tablet and one 100 mg ritonavir capsule at 7:00 a.m. after an overnight fast. A final dose of ritonavir was administered at 7:00 p.m. that evening.
Arm/Group | Colchicine Alone | Ritonavir Alone | Colchicine With Steady-state Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3 | 2 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Ritonavir Alone | Colchicine With Steady-state Ritonavir
upper abdominal pain (Gastrointestinal disorders) | 1/24 (1) | 0/18 (0) | 0/18 (0)
nausea (Gastrointestinal disorders) | 1/24 (1) | 0/18 (0) | 1/18 (1)
vomiting (Gastrointestinal disorders) | 1/24 (2) | 0/18 (0) | 0/18 (0)
gastroenteritis viral (Infections and infestations) | 1/24 (1) | 0/18 (0) | 0/18 (0)
dysgeusia (Nervous system disorders) | 1/24 (1) | 0/18 (0) | 1/18 (1)
headache (Nervous system disorders) | 1/24 (1) | 0/18 (0) | 1/18 (1)
dysmenorrhoea (Reproductive system and breast disorders) | 0/24 (0) | 0/18 (0) | 1/18 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/18 (1) | 0/18 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/18 (1) | 0/18 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2/24 (2) | 0/18 (0) | 0/18 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 2/18 (2) | 0/18 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days